CLINICAL TRIAL: NCT05142540
Title: Detection and Characterization of Anti-SARS-CoV-2 Salivary Antibodies After COVID-19 Booster Vaccines - The CoVVacBoost Study
Brief Title: Detection and Characterization of Anti-SARS-CoV-2 Salivary Antibodies After COVID-19 Booster Vaccines
Acronym: CoVVacBoost
Status: Terminated | Type: Observational
Why Stopped: No more booster vaccinations are being carried out at the site. Further recruitment is therefore not possible.
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: CoVVacBoost
Record Dates: First submitted 2021-12-01; First posted 2021-12-02 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Anti-SARS-CoV-2 Antibody Response
Keywords: Vaccination
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- blood and saliva sampling: blood and saliva samples will be taken
  Interventions: Procedure: blood and saliva samples will be taken

INTERVENTIONS:
Procedure: blood and saliva samples will be taken — For serology, 8 ml of blood and 1.5 ml saliva samples will be taken at every visit.
  For testing cellular immunity, additional 24 ml of blood will be drawn at visits 1 and 2.

SUMMARY:
The investigators aim to evaluate the ability of a COVID-19 (Coronavirus disease) booster vaccine to induce a salivary antibody response and investigate a possible correlation with the serum antibody response and the cellular response.

The investigators will conduct a prospective single center cohort study including fully vaccinated probands.

DETAILED DESCRIPTION:
The investigators will conduct a prospective single center cohort study including fully vaccinated probands.. The study will take place at the Medical University of Graz. Blood and saliva samples will be obtained before the third booster vaccination, 3-8 weeks, and 6 months after the third booster vaccination.

The total duration of the study is 15 months, starting in November 2021 with a recruiting period until June 2022 and termination of all scheduled visits until January 2023.

In order to be enrolled, participants must be 18 years or older, able to understand study procedures, provide written informed consent (Biobank informed consent and study specific informed consent).Scheduled vaccination for the booster vaccination with Comirnaty or Spikevax will allow recruitment.

At Visit 1, after informed consent, inclusion and exclusion criteria will be checked to include or exclude the subject in the trial. Clinical history will be assessed and blood (32ml - Serology, T cell immunity) and saliva (1.5ml) will be taken. At visit 2, 3-8 weeks after after 3rd vaccination, vaccination reactions and clinical history will be assessed. Blood (32ml - serology, T cell immunity) and saliva (1.5ml) will be taken.

At vist 3,6 Month (±3 weeks) after 3rd vaccination, clinical history will be assessed. Blood (8ml - serology) and saliva (1.5ml) will be taken.

Antibody tests and T cell assays will be performed according to protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Individuals who received full vaccination with any authorized COVID-19 vaccine and decided to receive a booster vaccination as recommended by national guidelines. -

Exclusion Criteria:

1. Presence of diseases or therapies that are likely to interfere with the immune response to booster vaccination.
2. Any contraindications to the vaccine planned to receive as listed in the product characteristics.
3. Lack of willingness to undergo serial blood draws and attend follow-up appointments.
4. Having already received a third (booster) vaccination with any COVID-19 vaccine.
5. Women who are pregnant or breastfeeding.
6. Persons who are not willing to sign the informed consents (biobank informed consent and study specific informed consent) -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Individuals who received full vaccination with any authorized COVID-19 vaccine
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Immunoglobulin (Ig)A concentrations to anti-SARS (severe acute respiratory syndrome)-CoV-2 spike protein in saliva. | 3-8 weeks after the third booster vaccination
  IgA concentrations to anti-SARS-CoV-2 spike protein in saliva before the third booster vaccination and 3-8 weeks after the third booster vaccination measured by SARS-CoV-2 antigen-binding Ig assays and life virus and pseudovirus neutralizing assays.
IgG concentrations to anti-SARS-CoV-2 spike protein in saliva. | 3-8 weeks after the third booster vaccination
  IgG concentrations to anti-SARS-CoV-2 spike protein in saliva before the third booster vaccination and 3-8 weeks after the third booster vaccination measured by SARS-CoV-2 antigen-binding Ig assays and life virus and pseudovirus neutralizing assays.
IgM concentrations to anti-SARS-CoV-2 spike protein in saliva. | 3-8 weeks after the third booster vaccination
  IgM concentrations to anti-SARS-CoV-2 spike protein in saliva before the third booster vaccination and 3-8 weeks after the third booster vaccination measured by SARS-CoV-2 antigen-binding Ig assays and life virus and pseudovirus neutralizing assays.

SECONDARY OUTCOMES:
IgA concentrations to anti-SARS-CoV-2 spike protein in serum | 3-8 weeks after the third booster vaccination
  IgA concentrations to anti-SARS-CoV-2 spike protein in serum before the third booster vaccination and 3-8 weeks after the third booster vaccination
IgG concentrations to anti-SARS-CoV-2 spike protein in serum | 3-8 weeks after the third booster vaccination
  IgG concentrations to anti-SARS-CoV-2 spike protein in serum before the third booster vaccination and 3-8 weeks after the third booster vaccination
IgM concentrations to anti-SARS-CoV-2 spike protein in serum | 3-8 weeks after the third booster vaccination
  IgM concentrations to anti-SARS-CoV-2 spike protein in serum before the third booster vaccination and 3-8 weeks after the third booster vaccination
IgA concentrations to anti-SARS-CoV-2 spike protein in saliva and serum | 3-8 weeks after the third booster vaccination
  IgA concentrations to anti-SARS-CoV-2 spike protein in saliva and serum before the third booster vaccination and 6 months after the third booster vaccination
IgG concentrations to anti-SARS-CoV-2 spike protein in saliva and serum | 3-8 weeks after the third booster vaccination
  IgG concentrations to anti-SARS-CoV-2 spike protein in saliva and serum before the third booster vaccination and 6 months after the third booster vaccination
IgM concentrations to anti-SARS-CoV-2 spike protein in saliva and serum | 3-8 weeks after the third booster vaccination
  IgM concentrations to anti-SARS-CoV-2 spike protein in saliva and serum before the third booster vaccination and 6 months after the third booster vaccination
Reactivity of T cells specific for recombinant S protein or other antigens of respiratory pathogens | 3-8 weeks after the third booster vaccination
  Reactivity of T cells specific for recombinant S protein or other antigens of respiratory pathogens including endemic coronaviruses before the third booster vaccination and 3-8 weeks and 6 months after the third booster vaccination.
Detection of antibodies against other respiratory pathogens | 3-8 weeks after the third booster vaccination
  Detection of antibodies against other respiratory pathogens including endemic coronaviruses which might be associated with the response to booster COVID-19 vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stradner, Principal Investigator — Medical University Graz Austria
Locations (1):
- Medizinische Universität Graz, Klinische Abteilung für Rheumatologie und Immunologie, Graz, Austria